CLINICAL TRIAL: NCT04577651
Title: Study to Evaluate Boston Scientific Vercise Cartesia 16-contact Directional Lead (X/HX) With Deep Brain Stimulation (DBS) Systems for the Treatment of Parkinson's Disease (PD)
Brief Title: Cartesia eXTend 3D Study
Acronym: eXTend 3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4092
Record Dates: First submitted 2020-09-26; First posted 2020-10-08 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- 16-contact Directional Deep Brain Stimulation (Experimental): Deep Brain Stimulation with a 16-contact Directional Lead
  Interventions: Device: 16-contact Directional Deep Brain Stimulation

INTERVENTIONS:
Device: 16-contact Directional Deep Brain Stimulation — Deep Brain Stimulation with 16-contact Directional Lead

SUMMARY:
The purpose of the study is to document patient outcomes including effectiveness for Boston Scientific Corporation's Vercise Cartesia 16-contact Directional Lead(s) (X/HX) with Deep Brain Stimulation (DBS) systems for the treatment of Parkinson's Disease (PD).

DETAILED DESCRIPTION:
Subjects will receive Deep Brain Stimulation with a 16-contact Directional Lead to treat their Parkinson's Disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Candidate for DBS implant in the treatment of Parkinson's disease
* Must be on stable anti-parkinsonian medications for 28 days prior to Informed Consent
* Persistent disabling Parkinson's disease symptoms such as dyskinesias, motor fluctuations, or disabling "off" periods despite optimal medical therapy
* Be willing and able to comply with all visits and study related procedures (e.g., using the remote control, charging system, etc.).

Key Exclusion Criteria:

* Any intracranial abnormality or medical condition that would contraindicate DBS surgery
* Have any significant psychiatric or cognitive condition likely to compromise the subject's ability to comply with requirements of the study protocol (e.g. bipolar, schizophrenia, mood disorder with psychotic features, cluster B personality disorders)
* Any current drug or alcohol abuse, as determined by the investigator
* Any history of recurrent or unprovoked seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2025-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (10):
- Germany (6):
  - University Berlin, Charite Virchow Standort, Wedding, Berlin
  - Uniklinik Koeln, Cologne
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - UMC St. Radboud, Nijmegen
- United Kingdom (2):
  - St. Georges Hospital, London
  - John Radcliffe Hospital, Oxford

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 16-contact Directional Deep Brain Stimulation
Started | 58
Completed | 45
Not Completed | 13
Not completed — Screen Failure | 7
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of the Intent-to-Treat Population
Arm/Group | 16-contact Directional Deep Brain Stimulation
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Netherlands | 17
  United Kingdom | 10
  Germany | 22
MDS-UPDRS-III score (meds off condition) [Mean (Standard Deviation); unit: units on a scale] — Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating (MDS-UPDRS) Part III. Range 0 - 108. Higher scores indicate worse function.
  units on a scale | 47.9 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Function
Description: Mean change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating (MDS-UPDRS) Part III scores from Baseline in meds off condition to 12 weeks post device-activation in stim on/meds off condition. Range 0 - 108. Higher scores indicate worse function.
Time Frame: 12 weeks post device-activation
Population: Intent to treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16-contact Directional Deep Brain Stimulation
Number analyzed (Participants) | 49
units on a scale | -19.9 (12.8)

2. Secondary Outcome: Change in Motor Function
Description: Mean change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating (MDS-UPDRS) Part III scores from Baseline (meds off) to 26 weeks post device-activation (stim on/meds off). Range 0 - 108. Higher scores indicate worse function.
Time Frame: 26 weeks post device-activation
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16-contact Directional Deep Brain Stimulation
Number analyzed (Participants) | 45
units on a scale | -21.4 (11.9)

3. Secondary Outcome: Change in Motor Function
Description: Mean change in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating (MDS-UPDRS) Part III scores from Baseline (meds off) to 52 weeks post device-activation (stim on/meds off). Range 0 - 108. Higher scores indicate worse function.
Time Frame: 52 weeks post device-activation
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 16-contact Directional Deep Brain Stimulation
Number analyzed (Participants) | 41
score on a scale | -21.2 (14.0)

4. Secondary Outcome: Change in Quality of Life
Description: Mean change in Parkinson's Disease Questionnaire (PDQ-39) summary scores from Baseline (meds on) to 12 weeks post device-activation (stim on/meds on). Scores range from 0 to 100, with 0 representing perfect health and 100 representing worst health.
Time Frame: 12 weeks post device-activation
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16-contact Directional Deep Brain Stimulation
Number analyzed (Participants) | 48
units on a scale | -6.1 (11.0)

5. Secondary Outcome: Change in Quality of Life
Description: Mean change in Parkinson's Disease Questionnaire (PDQ-39) summary scores from Baseline (meds on) to 26 weeks post device-activation (stim on/meds on). Scores range from 0 to 100, with 0 representing perfect health and 100 representing worst health.
Time Frame: 26 weeks post device-activation
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16-contact Directional Deep Brain Stimulation
Number analyzed (Participants) | 46
units on a scale | -5.3 (11.4)

6. Secondary Outcome: Change in Quality of Life
Description: Mean change in Parkinson's Disease Questionnaire (PDQ-39) summary scores from Baseline (meds on) to 52 weeks post device-activation (stim on/meds on). Scores range from 0 to 100, with 0 representing perfect health and 100 representing worst health.
Time Frame: 52 weeks post device-activation
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16-contact Directional Deep Brain Stimulation
Number analyzed (Participants) | 42
units on a scale | -6.4 (11.5)

ADVERSE EVENTS:
Time Frame: Adverse Event Rates for all Subjects through the week 52 visit, approximately 14 months post informed consent.
Arm/Group | 16-contact Directional Deep Brain Stimulation
All-Cause Mortality (participants affected / at risk) | 1/58
Serious Adverse Events (participants affected / at risk) | 14/58
Other Adverse Events (participants affected / at risk) | 25/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 16-contact Directional Deep Brain Stimulation (N=58)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Implant site paraesthesia (General disorders) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 2 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 1 (1)
Fine motor skill dysfunction (Nervous system disorders) | 1 (1)
Hyperkinesia (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Dopamine dysregulation syndrome (Psychiatric disorders) | 1 (1)
Impulse-control disorder (Psychiatric disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 16-contact Directional Deep Brain Stimulation (N=58)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Parkinson's disease (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 4 (4)
Dyskinesia (Nervous system disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 4 (8)
Implant site pain (General disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT04577651/Prot_SAP_001.pdf